CLINICAL TRIAL: NCT02264184
Title: An Open Label Randomized Two-way Crossover Study to Investigate the Effect of Paroxetine Mediated CYP2D6 Inhibition on the Single Oral Dose Pharmacokinetics of Tamsulosin in Healthy Male Volunteers (CYP2D6 Extensive Metabolizers)
Brief Title: Study to Investigate the Effect of Paroxetine Mediated CYP2D6 Inhibition on the Pharmacokinetics of Tamsulosin in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 527.79
Record Dates: First submitted 2014-10-14; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Tamsulosin; AlnA protein, Acinetobacter radioresistens; Paroxetine

ARMS (2):
- Tamsulosin + Paroxetine (Experimental): Tamsulosin: q.d on day 1
  Paroxetine: higher dose q.d. on days -7 to 2 q.d., lower dose on days -10 to -8 and 3 to 5
  Interventions: Drug: Tamsulosin; Drug: Paroxetine
- Tamsulosin (Active Comparator): Tamsulosin: q.d on day 1
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Tamsulosin
  Other Names: Alna®
Drug: Paroxetine
  Other Names: Tagonis®
  Arms: Tamsulosin + Paroxetine

SUMMARY:
Study to investigate the effect of CYP2D6 inhibition by paroxetine on the single oral dose pharmacokinetics of tamsulosin and to investigate the effect on safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

All participants in the study are

* Healthy males
* Ranging from 21 to 50 years of age
* Body mass index (BMI) within 18.5 to 29.9 kg/m2
* In accordance with Good Clinical Practice (GCP) and the local legislation all volunteers will have given their written informed consent prior to admission to the study

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders, clinically relevant electrolyte disturbances
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or clinically relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24:00 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study or during the study
* Use of any drugs which might influence the results of the trial up to 7 days prior to enrolment in the study or during the study
* Participation in another trial with an investigational drug (within two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars of > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (> 100 mL within four weeks prior to administration or during the trial)
* Any laboratory value outside the reference range if indicative of underlying disease or poor health
* Excessive physical activities within the last week before the trial or during the trial
* Hypersensitivity to treatment medication and/or related drugs of these classes
* Non extensive metabolizer (EM) for CYP2D6

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum measured concentration of tamsulosin HCl in plasma) | up to 48 hours after dosing
AUC0-∞ (area under the concentration-time curve of tamsulosin HCl in plasma over the time interval from 0 extrapolated to infinity) | up to 48 hours after dosing

SECONDARY OUTCOMES:
tmax (time from dosing to the maximum measured concentration of tamsulosin HCl in plasma) | up to 48 hours after dosing
AUC0-tz (area under the concentration-time curve of tamsulosin HCl in plasma over the time interval from 0 to the last quantifiable data point) | up to 48 hours after dosing
λz (terminal rate constant of tamsulosin HCl in plasma) | up to 48 hours after dosing
t1/2 (terminal half-life of tamsulosin HCl in plasma) | up to 48 hours after dosing
MRTpo (mean residence time of tamsulosin HCl in the body after oral administration) | up to 48 hours after dosing
CL/F (apparent clearance of tamsulosin HCl in plasma after an extravascular administration) | up to 48 hours after dosing
Vz/F (apparent volume of distribution of tamsulosin HCl during the terminal phase λz following an extravascular administration) | up to 48 hours after dosing
RCmax,T/R (ratio of the Cmax value of the test treatment to the Cmax value of the reference treatment after single dose) | up to 48 hours after dosing
RAUC0-∞,T/R (ratio of the test treatment versus the reference treatment from zero to infinity, expressed as ratio of AUC values after single dose) | up to 48 hours after dosing
Number of subjects with adverse events | up to 21 days after last treatment
Assessment of tolerability by investigator on a 4-point scale | within 21 days after last treatment